CLINICAL TRIAL: NCT03464279
Title: Use of a Behavioral Economic Intervention to Reduce Antibiotic Prescription for Upper Respiratory Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: LAC+USC Medical Center (Other); Los Angeles County Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Catherine A. Sarkisian, Professor in Residence, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB #16-000932-004
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Antibiotics; Upper Respiratory Infections; Safety-Net Hospitals; Behavioral Economics; Choosing Wisely
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Site (Experimental): The intervention Site (Urgent Care Center at LAC+USC Medical Center) will receive a three part intervention consisting of (1) Email Choosing Wisely® guidelines and presented journal club to all 16 urgent care clinicians, (2) leveraging EHR performance data to provide individual clinicians with case-specific audit-feedback (both via emails and in-person while precepting nurse practitioners) on low-value antibiotic prescribing, and (3) using a behavioral "nudge", urgent care clinicians will sign a large poster committing to avoid prescribing low-value antibiotics for uncomplicated URIs displayed in the clinic.
  Interventions: Behavioral: Nudge using Behavioral Economic Interventions
- Control Site (Active Comparator): The control site (Urgent Care Center at Olive View-Medical Center) will receive broader health system efforts to reduce antibiotic prescribing consisting of Center for Disease Control prescription pads for non-antibiotic treatments (e.g., decongestants) that offer patients alternatives to antibiotics.
  Interventions: Behavioral: Standard Practices to Reduce Health System Antibiotic Prescription

INTERVENTIONS:
Behavioral: Nudge using Behavioral Economic Interventions
  Arms: Intervention Site
Behavioral: Standard Practices to Reduce Health System Antibiotic Prescription
  Arms: Control Site

SUMMARY:
In an effort to implement Choosing Wisely guidelines and decrease patient harm, we will implement and evaluate a clinician audit-feedback and behavioral "nudge" initiative to reduce low-value antibiotics for URIs. Using a quasi-experiment (pre-post) design, antibiotic prescriptions for URI at LAC+USC Urgent Care Center (intervention site) vs. Olive View-UCLA Urgent Care Center (control site) will used to test the effects of behavioral "nudge" on antibiotic prescribing.

DETAILED DESCRIPTION:
National prescription rates for low-value antibiotics for uncomplicated upper respiratory infections (URIs) remain unacceptably high, including at LAC+USC Medical Center-one of the largest safety net medical centers in the U.S. Using a quasi-experiment (pre-post) design, antibiotic prescriptions for URI at LAC+USC Urgent Care Center (intervention site) vs. Olive View-UCLA Urgent Care Center (control site) will be compared. A three-part intervention at LAC+USC consists of (1) the urgent care medical director emailing Choosing Wisely® guidelines and presented journal club to all 16 urgent care clinicians, and then (2) leveraging EHR performance data to provide individual clinicians with case-specific audit-feedback (both via emails and in-person while precepting nurse practitioners) on low-value antibiotic prescribing, and (3) using a behavioral "nudge", urgent care clinicians will sign a large poster committing to avoid prescribing low-value antibiotics for uncomplicated URIs, which will be displayed in the clinic. In contrast, the control site (Urgent Care Center at Olive View-Medical Center) will receive Centers for Disease Control prescription pads for non-antibiotic treatments (e.g., decongestants) that offer patients alternatives to antibiotics, in a broader health system effort to reduce antibiotic prescribing. Patient with URIs (e.g., acute bronchitis, bronchitis NOS, excluding guideline-based red flags such as COPD, HIV) will be identified using electronic health record clinical billable data and low-value antibiotic prescriptions rates per visit will be monitored at both sites. Differences in prescriptions rates will be determined using an interrupted time-series analysis comparing utilization between sites using a repeated measures logistic regression model.

.

ELIGIBILITY:
Inclusion Criteria:

* all patient receiving treatment for Upper Respiratory Infections (defined by ICD codes EHR billable codes) at both LAC+USC Medical Center Urgent Care or Olive View-UCLA Medical Center

Exclusion Criteria:

* Patients not receiving treatment for Upper Respiratory Infections at both LAC+USC Medical Center Urgent Care or Olive View-UCLA Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Low-value antibiotic prescriptions rates per visit | 1 year
  Changes in inappropriate antibiotic prescriptions rates per visit before and after implementation of intervention at both sites

SECONDARY OUTCOMES:
Coding Shift (ie, a shift in use of diagnostic codes to conditions that are more antibiotic appropriate) in URI diagnosis | 1 year
  Change frequency of proportion of antibiotic appropriate diagnoses before intervention and after at both sites.

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles County +University of Southern California (LAC+USC) Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Meeker D, Knight TK, Friedberg MW, Linder JA, Goldstein NJ, Fox CR, Rothfeld A, Diaz G, Doctor JN. Nudging guideline-concordant antibiotic prescribing: a randomized clinical trial. JAMA Intern Med. 2014 Mar;174(3):425-31. doi: 10.1001/jamainternmed.2013.14191. PMID 24474434
- [Background] Gonzales R, Steiner JF, Lum A, Barrett PH Jr. Decreasing antibiotic use in ambulatory practice: impact of a multidimensional intervention on the treatment of uncomplicated acute bronchitis in adults. JAMA. 1999 Apr 28;281(16):1512-9. doi: 10.1001/jama.281.16.1512. PMID 10227321